CLINICAL TRIAL: NCT04388683
Title: Prevention of COVID-19 Progression Through Early Administration of Inhaled Nitric Oxide.
Brief Title: Inhaled Nitric Oxide for Preventing Progression in COVID-19
Acronym: NO-COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Bellerophon requested study to be stopped.
Sponsor: Tufts Medical Center (Other)
Collaborators: Bellerophon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000554
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19; Inhaled Nitric Oxide
MeSH Terms: conditions — COVID-19 | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive study drug treatment.
  Interventions: Drug: Nitric Oxide
- Control (No Intervention): Will receive standard of care.

INTERVENTIONS:
Drug: Nitric Oxide — Subjects will receive iNO using the INO pulse device at a dose of 125 mcg/kg IBW/hr (equivalent to approximately 20 ppm). The clinical disease severity will be assessed pre-randomization as the worse of 2 scores measured 2 hours apart. Patients eligible for randomization will be those with scores of 1 or 2 (below), and randomization will be stratified according to score (1 or 2). Study drug will begin within 1 hour of randomization. Beginning on the day following randomization ("day 1"), we will be calculate clinical score, daily, as the average of 3 measurements taken within 2 hour windows centered at 6AM, 2PM, and 10PM.
  Arms: Intervention

SUMMARY:
This is a pilot randomized-controlled (2:1) open label investigation of inhaled NO to prevent progression to more advanced disease in 42 hospitalized patients with COVID-19, at risk for worsening, based on baseline systemic oxygenation and 2 or more of the major risk factors of age > 60 years, type II DM, hypertension, and obesity.

DETAILED DESCRIPTION:
Primary Objective:

• To investigate the hypothesis that inhaled NO will reduce clinical worsening of hospitalized, high-risk patients with early COVID-19 to progressive systemic de-oxygenation, intubation, or death.

Secondary Objectives:

• To investigate the hypothesis that the beneficial effects of inhaled NO occur coincident with a decrease in systemic inflammation in COVID-19.

This is a pilot randomized-controlled (2:1) open label investigation of inhaled NO to prevent progression to more advanced disease in 42 hospitalized patients with COVID-19, at risk for worsening, based on baseline systemic oxygenation and 2 or more of the major risk factors of age > 60 years, type II DM, hypertension, and obesity.

We will perform computerized block randomization (on day zero) with a 2:1 study drug-to-control ratio to receive either open label pulsed inhaled nitric oxide, in addition to standard of care, or standard of care alone. Randomization will be stratified by being in clinical severity stage 1 or stage 2. Randomization will occur in blocks of 6 subjects: 4 iNO and 2 standard of care. Subjects will receive iNO using the INO pulse device at a dose of 125 mcg/kg IBW/hr (equivalent to approximately 20 ppm)

The clinical disease severity will be assessed pre-randomization as the worse of 2 scores measured 2 hours apart. Patients eligible for randomization will be those with scores of 1 or 2 (below), and randomization will be stratified according to score (1 or 2). Study drug will begin within 1 hour of randomization. Beginning on the day following randomization ("day 1"), we will be calculate clinical score, daily, as the average of 3 assessments made within 2 hour windows.

The patient will be followed, and clinical stage determined daily, through discharge, death or 28 days post-randomization. Treatment will be given for up to 2 weeks unless patient deteriorates and requires escalation to high flow or intubation or improves and is no longer deemed to need therapy.

The following severity score 3 times daily, based on the level of oxygenation / ventilation support, where the treatment target is 92% <= O2 saturation < 96%

: Scale Title:7-Point Respiratory Severity Scale Scale Range: 0-6 Higher values = worse

Stage Oxygen support

0. Not receiving O2 supplementation; AND room air O2 saturation ≥95%

1. Supplemental O2 ≤ 2 liters/min; OR room air O2 saturation ≤ 94%
2. Supplemental nasal O2 >2 and <= 5 liters/min
3. Supplemental nasal O2 >5 liters/min
4. HFNC or NIV with FiO2 > 50%
5. Intubation, ECMO, or need to intubate with "Do not intubate" order
6. Death

Treatment effect will also be assessed, as a secondary endpoint, via an alternate severity scale, assigned daily from the data accrued, as above, through 14 days post-randomization or discharge.

Data from this pilot study will be used to plan future a larger randomized controlled outcome trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years.
2. Admitted to the hospital (med-surg or critical care) with dyspnea
3. Diagnosis of COVID-19 based on either

   1. positive nasal or oral pharyngeal swab by PCR, or
   2. highly probable clinical picture based on clinical and CXR/CT scan
4. Requiring oxygen supplementation OR O2 saturation on room air of ≤ 94%
5. At least 2 of the following 4 risk factors for clinical worsening:

   1. Age >= 60 years
   2. T2DM or pre-diabetes as evidenced by either treatment with a hypoglycemic agent or any documented HgA1c >= 5.6
   3. Obesity, based on BMI >= 30 kg/m2
   4. Hypertension, based on treatment with an antihypertensive medication or systolic or diastolic blood pressure measurement >= 140 or >= 90 mmHg, documented at enrollment or at any time within the prior 6 months.

Exclusion Criteria:

1. Intubated or prior intubation (during present hospitalization) or anticipated intubation within the subsequent 2 hours.
2. Receiving > 5L/min flow nasal O2 to maintain O2sat greater than or equal to 92%
3. Using high-flow nasal cannula (HFNC) or non-invasive ventilation (NIV)
4. Receiving iNO, a PDE5 inhibitor, oral or intravenous nitrates, nitroprusside, prilocaine, sulfonamides, or riociguat.
5. Other major pulmonary, cardiac, such as chronic obstructive lung disease or heart failure, or systemic illness or disease involvement with potential to represent the primary driver for clinical deterioration within the next 3 days.
6. History of group 1 pulmonary hypertension.
7. Pregnancy
8. Active breast feeding
9. Severe chronic kidney disease, either receiving renal replacement therapy or eGFR < 15 ml/min/m2
10. Acute kidney injury (AKI), evidenced by acute doubling of serum creatinine within previous 48 hours.
11. Clinically relevant spontaneous alteration of mental state
12. Inability to provide written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Konstam, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data from this pilot study will be used to plan future a larger randomized controlled outcome trial.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that 9 participants signed consent forms. However, only 8 participants completed the study because the last patient was consented the morning the study was shut down, so they did complete treatment steps or have data collected for them.
Groups:
- Inhaled Nitric Oxide: Will receive study drug treatment.
  Nitric Oxide: Subjects will receive iNO using the INO pulse device at a dose of 125 mcg/kg IBW/hr (equivalent to approximately 20 ppm). The clinical disease severity will be assessed pre-randomization as the worse of 2 scores measured 2 hours apart. Patients eligible for randomization will be those with scores of 1 or 2 (below), and randomization will be stratified according to score (1 or 2). Study drug will begin within 1 hour of randomization. Beginning on the day following randomization ("day 1"), we will be calculate clinical score, daily, as the average of 3 measurements taken within 2 hour windows centered at 6AM, 2PM, and 10PM.
- Standard of Care: Will receive standard of care.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Standard of Care
Started | 6 | 3
Completed | 5 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (14.2) | 46.7 (1.5) | 58.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9
Clinical Disease Severity Score [Count of Participants; unit: Participants] — The clinical disease severity will be assessed pre-randomization as the worse of 2 scores measured 2 hours apart. Patients eligible for randomization will be those with scores of 1 or 2. Stages are defined below.
  Stage Oxygen support 0 Not receiving O2 supplementation; AND room air O2 saturation ≥95%
  1. Supplemental O2 ≤ 2 liters/min; OR room air O2 saturation ≤ 94%
  2. Supplemental nasal O2 >2 and ≤ 5 liters/min
  3. Supplemental nasal O2 >5 liters/min
  4. HFNC or NIV with FiO2 > 50%
  5. Intubation, ECMO, or need to intubate with "Do not intubate" order
  6. Death
  Participants
    Stage 1 | 5 | 2 | 7
    Stage 2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Average Maximum Disease Severity Assessed Through 28 Days
Description: The clinical disease severity was assessed pre-randomization as the worse of 2 scores measured 2 hours apart. Patients eligible for randomization were those with scores of 1 or 2 (below), and randomization was stratified according to score (1 or 2). Study drug began within 1 hour of randomization. Beginning on the day following randomization ("day 1"), we calculated clinical score, daily, as the average of 3 measurements taken within 2 hour windows centered at 6AM, 2PM, and 10PM.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Participants
  Max. Clinical Disease Severity Score : Not receiving O2 Supp.; AND room air O2 saturation >95% | 1 | 1
  Max. Clinical Disease Severity Score : Supplemental O2 ≤2 liters/min; OR room air O2 saturation ≤94% | 3 | 1
  Max. Clinical Disease Severity Score : Supplemental nasal O2 >2 & ≤5 liters/min | 1 | 0
  Max. Clinical Disease Severity Score : HFNC or NIV with FiO2 >50% | 0 | 1
  HFNC or NIV with FiO2 >50% | 0 | 1

2. Secondary Outcome: Days to Maximum Clinical Disease Severity Score
Description: The number of days for participants to reach their maximum clinical disease severity score. Severity score assessed by the following table Stage Oxygen support 0 Not receiving O2 supplementation; AND room air O2 saturation ≥95%
  1. Supplemental O2 ≤ 2 liters/min; OR room air O2 saturation ≤ 94%
  2. Supplemental nasal O2 >2 and ≤ 5 liters/min
  3. Supplemental nasal O2 >5 liters/min
  4. HFNC or NIV with FiO2 > 50%
  5. Intubation, ECMO, or need to intubate with "Do not intubate" order
  6. Death
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Days | 1.0 [1.0 to 1.0] | 1 [1.0 to 2.0]

3. Secondary Outcome: Days to Maximum Outcome Severity Score
Description: The number of days for patients to reach maximum severity score from randomization. clinical score, daily, as the average of 3 measurements taken within 2 hour windows centered at 6AM, 2PM, and 10PM according to the following table:
  The following severity score 3 times daily, based on the level of oxygenation / ventilation support, where the treatment target is 92% ≤ O2 saturation < 96%:
  Stage Oxygen support 0 Not receiving O2 supplementation; AND room air O2 saturation ≥95%
  1. Supplemental O2 ≤ 2 liters/min; OR room air O2 saturation ≤ 94%
  2. Supplemental nasal O2 >2 and ≤ 5 liters/min
  3. Supplemental nasal O2 >5 liters/min
  4. HFNC or NIV with FiO2 > 50%
  5. Intubation, ECMO, or need to intubate with "Do not intubate" order
  6. Death HFNC = high-flow nasal cannula; NIV = non-invasive ventilation
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Days | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 8.0]

4. Secondary Outcome: Number of Participants in Each Stage at Maximum Severity
Description: Maximum outcome severity score
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Participants
  Hospitalized, requiring supp. O2 | 1 | 1
  Hospitalized, not requiring supp. O2 or ongoing medical care | 3 | 2
  Not hospitalized, no limitations on activities | 1 | 0

5. Secondary Outcome: Length of Hospital Stay
Description: The numbers of days a patient spent in the hospital.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Days | 3.0 [3.0 to 9.0] | 3.0 [2.0 to 5.0]

6. Secondary Outcome: Mortality
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were monitored for up to 28 days after randomization.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

LIMITATIONS AND CAVEATS:
The study was terminated early by request of the company providing the iNO Drug. Our data set is small are analysis was effected by this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT04388683/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04388683/ICF_001.pdf